CLINICAL TRIAL: NCT01257997
Title: Quantification of Human Adipogenesis
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Matthew Steinhauser, MD, Attending Physician, Brigham and Women's Hospital
Other Study IDs: BWH-2010p001900
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: No specific experimental conditions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fat biopsy. Oral mucosal smear. White blood cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy subjects: 18-49 year old healthy men and women. Free of significant chronic medical illness and illicit substance abuse. Body mass index from 20 to 27.
  Interventions: Biological: 15N-Thymidine, 2H-Water

INTERVENTIONS:
Biological: 15N-Thymidine, 2H-Water — Stable isotope 15N-thymidine, infused IV (15mg/hour) for 72 hours (phase 1 pilot).
  Stable isotope 2H-water, ingested by mouth once per day for 3 days (phase 1 pilot) or 28 days (phase 2 pilot).

SUMMARY:
This pilot study is using a novel technology to measure the rate of turnover of new fat cells. Analysis of volunteer samples is ongoing, however the study is currently not enrolling new volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-49 years.
* Healthy.

Exclusion Criteria:

* Significant chronic medical illness.
* Illicit substance or alcohol abuse.
* Body mass index > 27 kg/meters squared.
* Underweight (BMI < 20 kg/m2).
* History of keloid formation (excessive scarring).
* Pregnant.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers. Aged 18-49 years. Free of significant chronic medical illness. Free of illicit substance abuse.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-12; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Quantifying human adipogenesis-counting the number of new fat cells. | 4 weeks-7 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Steinhauser, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Steinhauser ML, Bailey AP, Senyo SE, Guillermier C, Perlstein TS, Gould AP, Lee RT, Lechene CP. Multi-isotope imaging mass spectrometry quantifies stem cell division and metabolism. Nature. 2012 Jan 15;481(7382):516-9. doi: 10.1038/nature10734. PMID 22246326